CLINICAL TRIAL: NCT05461274
Title: An In Depth Study Examining Patterns in the Clinical Trial Experiences of Diabetic Neuropathy Patients
Brief Title: Determining Patterns In Trial Experiences of Diabetic Neuropathy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 8874740
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Neuropathies; Diabetic Neuropathy Peripheral
Keywords: diabetic neuropathy; neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical studies is highly skewed towards particular demographic groups of people.

This study will invite several participants to gather a wide range of information on clinical trial experiences for diabetic neuropathy patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of diabetic neuropathy.

The data collected from this study will help improve future outcomes for all diabetic neuropathy patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient plans to participate in an interventional clinical trial for the condition of diabetic neuropathy
* Patient has been diagnosed with a type of diabetic neuropathy
* Patient is a minimum of 18 years of age
* Patient has access to a home internet connection in order to provide regular updates through the course of the study

Exclusion Criteria:

* Patient is not able to provide consistent digital updates as per study requirements
* Patient does not complete or agree to terms outlined in the Informed Consent Form
* Patient has an ECOG score of 4 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic neuropathy who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an diabetic neuropathy clinical trial | 3 months
Rate of patients who remain in diabetic neuropathy clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clark LT, Watkins L, Pina IL, Elmer M, Akinboboye O, Gorham M, Jamerson B, McCullough C, Pierre C, Polis AB, Puckrein G, Regnante JM. Increasing Diversity in Clinical Trials: Overcoming Critical Barriers. Curr Probl Cardiol. 2019 May;44(5):148-172. doi: 10.1016/j.cpcardiol.2018.11.002. Epub 2018 Nov 9. PMID 30545650
- [Background] Pfeifer MA, Schumer MP. Clinical trials of diabetic neuropathy: past, present, and future. Diabetes. 1995 Dec;44(12):1355-61. doi: 10.2337/diab.44.12.1355. PMID 7589838
- [Background] Rosenberger DC, Blechschmidt V, Timmerman H, Wolff A, Treede RD. Challenges of neuropathic pain: focus on diabetic neuropathy. J Neural Transm (Vienna). 2020 Apr;127(4):589-624. doi: 10.1007/s00702-020-02145-7. Epub 2020 Feb 8. PMID 32036431

DOCUMENTS (1):
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT05461274/ICF_000.pdf